CLINICAL TRIAL: NCT03737344
Title: Phase II Trial of Interleukin-1 Receptor Antagonist in Intracerebral Haemorrhage: BLOcking the Cytokine IL-1 in ICH
Brief Title: BLOC-ICH: Interleukin-1 Receptor Antagonist in Intracerebral Haemorrhage
Acronym: BLOC-ICH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adrian Parry-Jones (Other)
Collaborators: Northern Care Alliance NHS Foundation Trust (Other); National Institute for Health Research, United Kingdom (Other Government); Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor-Investigator, Adrian Parry-Jones, NIHR Clinician Scientist & Honorary Consultant Neurologist, University of Manchester
Organization: University of Manchester (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R118439
Record Dates: First submitted 2018-10-18; First posted 2018-11-09 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Intracerebral Haemorrhage
Keywords: haemorrhage; Stroke; Bleeding
MeSH Terms: conditions — Cerebral Hemorrhage; Hemorrhage; Stroke | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IL-1Ra Kineret® (Active Comparator): 100mg doses of the trial drug Kineret® will be administered subcutaneously (SC) twice daily (12 hourly) starting within 8 hours of symptoms onset for a maximum of 3 days from symptoms onset (or sooner if discharged from neurosurgical centre).
  Interventions: Drug: IL-1Ra Kineret®
- IL-1Ra Placebo (Placebo Comparator): 100mg doses of the placebo will be administered subcutaneously (SC) twice daily (12 hourly) starting within 8 hours of symptoms onset for a maximum of 3 days from symptoms onset (or sooner if discharged from neurosurgical centre).
  Interventions: Other: IL-1Ra Placebo

INTERVENTIONS:
Drug: IL-1Ra Kineret® — Kineret® 100 mg in 0.67 ml Prefilled Syringe
  Other Names: Anakinra
  Arms: IL-1Ra Kineret®
Other: IL-1Ra Placebo — Placebo identical to Kineret® 100 mg in 0.67 ml Prefilled Syringe
  Arms: IL-1Ra Placebo

SUMMARY:
This trial will help inform the development of a new treatment for intracerebral haemorrhage (ICH; also known as haemorrhagic stroke). ICH is a type of stroke caused by spontaneous bleeding into the brain. In the hours to days after bleeding occurs, inflammation develops in the brain around the haematoma (collection of blood in the brain). Inflammation is the body's natural response to injury, however when it continues unchecked there is a risk that the brain tissue around the haematoma will become swollen. This type of swelling can worsen existing stroke symptoms or cause new deficits such as speech disturbance and limb weakness, which can lead to long term disability.

The level of inflammation in the blood is high after ICH. The investigators want to investigate whether blocking this inflammation can improve overall recovery. The investigators research group has extensively investigated the use of a well-established anti-inflammatory drug, Kineret® in trials with patients who have suffered a stroke or brain haemorrhage. Kineret® is similar to a naturally-produced protein called interleukin-1 receptor antagonist (IL-1Ra) and is already licensed to treat patients with rheumatoid arthritis. The investigators have evidence from these previous studies that Kineret® reduced levels of inflammation in the blood after ischaemic stroke (caused by a blockage in an artery). However, in order to develop Kineret® as a treatment for ICH, the investigators need to know if it reduces levels of inflammation present in the blood following ICH and if it reduces swelling in the brain.

DETAILED DESCRIPTION:
The investigators know from previous studies that the level of inflammation in the blood is high after haemorrhagic stroke and want to investigate whether blocking this inflammation can improve outcomes. The only current treatments for haemorrhagic stroke are aimed at significantly reducing the blood pressure and reversing the action of any anticoagulants (e.g. warfarin) where necessary. Surgery to remove the blood clot is not an option for all participants and the benefits of this are not clear.

The investigators research group has extensively investigated the use of a well-established anti-inflammatory drug, Kineret® in trials with participants who have suffered a stroke or brain haemorrhage. Kineret® is similar to a naturally-produced protein called interleukin-1 receptor antagonist (IL-1Ra) and is already licensed to treat patients with rheumatoid arthritis. The investigators have evidence from these previous studies that Kineret® reduced levels of inflammation in the blood after ischaemic stroke (caused by a blockage in an artery). In another trial, the investigators collected samples of the haematoma blot clot removed during surgery in 47 participants who had suffered a haemorrhagic stroke. These participants were taking part in a trial of 'keyhole' surgery as a treatment for haemorrhagic stroke. The investigators found that higher levels of naturally occurring IL-1Ra in and around the haematoma blood clot is linked to less brain swelling a few days later. This suggests that Kineret® may reduce swelling in the brain after haemorrhagic stroke. However, in order to develop Kineret® as a treatment for haemorrhagic stroke, the investigators need to know if it reduces levels of inflammation present in the blood and if it reduces swelling in the brain.

The investigators also want to investigate whether blocking inflammation can improve outcomes following ICH. If the results of this trial show promise, it could support the decision to run a much larger trial to establish whether lowering inflammation improves recovery after haemorrhagic stroke.

Patients admitted to a neurosurgical centre within 8 hours of intracerebral haemorrhage (ICH) on brain imaging will be considered for study participation. Potential participants will be identified by the clinical team and will be referred to the research teams at the sites following usual and established pathways. These pathways may include potential participants being identified by; (i) Screening the acute referral databases/medical records, (ii) Attendance at ward round and, (iii) Referral by Accident and Emergency team. All members of the research teams at the sites have an existing working relationship with the clinical teams and are employed by the research site (hospital Trust). This procedure is employed at sites in order to identify potential participants for all acute and hyper acute research studies.

Capacity to consent may be an issue within this patient group. An appropriately trained member of the research team will carry out a formal assessment of capacity, where appropriate. Where it is not possible to obtain consent from the patient due to lack of capacity, the investigators will seek consent from their personal legal representative. If the patient lacks capacity to consent to participation and no personal legal representative exists, the decision to include the patient will be made by a senior member of the clinical team who is independent of the research team (professional legal representative).

In the event that a patient has the capacity to consent to participation, but is unable to complete and sign the relevant consent form due to physical difficulties resulting from their clinical condition or pre-existing physical impairments (e.g. visual difficulties or limb weaknesses), witnessed, verbal consent will be obtained. The patient will be asked to orally confirm their willingness to participate in each stage of the trial to the professional legal representative (most likely a member of the clinical team independent of the research group) who will then be asked to confirm this consent in writing. In the event that the physical difficulties resolve during the patient's inclusion in the trial, a further consent form will be completed.

Where initial consent is obtained from the patient's personal legal representative or the professional legal representative, the capacity of the patient to consent will be reassessed before each research assessment/intervention. If the patient regains capacity, they will be given information about the trial and asked to confirm willingness to continue trial participation by signing a consent form. Where initial consent is given by the patient, it will be made clear that they will remain in the trial should capacity be lost unless the decision to withdraw them is made by their representative, the research team, or by their clinical team.

Consent to trial participation will include sharing of personal contact data with the trial centre in order to conduct follow up assessment and the optional consent to storage of blood samples for use in other ethically-approved research.

Following consent, the research nurse will conduct an initial 'baseline' assessment. This will be written in the medical notes and also in an individual research file (Case Report Form). This first assessment will record details of how well the patient was at the time of inclusion in the trial as well as how well they were in the 3 months before stroke. The assessment will also record information such as age, sex and ethnicity and past medical history (including recent infections, previous stroke, risk factors, medications and vaccinations). A physical examination will record measurements of temperature, heart rate and blood pressure. A similar assessment will be repeated on each of the following 4 days after symptom-onset. The final assessment will be completed the morning after the final injection has been given. After this assessment the research team will ask the patient to verbally reconfirm consent that contact details can be passed to the coordinating centre (Chief Investigator's Team at University of Manchester) In addition to the baseline assessment, a research blood sample will be obtained to measure levels of inflammation at baseline. This blood sample will be up to 10ml (2 teaspoons) and will be taken from existing venous lines (where possible) to minimise discomfort for the participant.

After obtaining the baseline blood samples and baseline assessments, the participant will be randomised to treatment arm or placebo. The system will generate a unique participant identification number which will be used on all documentation from this point to identify subsequent samples, for communications and for data collection purposes. First dose of trial medication must be delivered within 8 hours of ICH and as soon as possible after randomisation.

Participants will receive 6 injections of identical doses of Trial Drug (Kineret® or placebo) over 3 days after ICH. However, only half the participants will receive Kineret® and the other half will receive placebo (dummy drug). The investigators will measure and compare levels of inflammation in the blood of both groups of participants before and after treatment with Trial Drug to assess if inflammation is lower in those who receive Kineret® compared to those given placebo. The investigators will also assess all brain imaging performed on trial participants in both treatment groups during their in-patient stay to see if there are differences in the number showing signs of further bleeding and brain swelling. If the results of this trial show promise, it could support the decision to run a much larger trial to establish whether lowering inflammation improves recovery after ICH.

At approximately 3 days after randomisation, the patient will undergo a repeat CT brain scan as part of the research trial. This scan is the same type as the one performed at admission. Although this scan is being performed as part of the research trial, the results will also be available to the doctors looking after the patient and may assist them in deciding on specific treatments. This scan will take approximately 10 minutes to perform but the participant may be away from the ward or department for up to 45 minutes. The scan will be used by the researchers who will compare it to brain imaging performed on admission to hospital.

In addition to the CT scan, participants may also be asked to undergo a Magnetic Resonance (MR) brain scan between 2-4 days from the onset of the stroke symptoms. This is optional and is dependent on availability of hospital scan appointments. Members of the research team at the recruiting hospital will record everything that happens to the patient during their in-patient stay. At 30 days after randomisation, participants will be followed up to further check their well-being. If the patient is still in hospital on this date, this assessment may be performed face-to-face by a member of the research team. However, if the participant has been discharged home or returned to their local hospital, the researcher will perform this assessment by telephone with the participant or their relative/friend if they are not able or their local healthcare provider. It is expected that this assessment will take around 45 minutes.

The participant will be contacted again by telephone at approximately 90 days (3 months) by a member of the research team at the trial coordinating centre in Manchester. This assessment will assess the participant's recovery after ICH and will include questions about their mood, level of fatigue and quality of life. It is expected that this assessment will take around 45 minutes. If for any reason, the participant is unable to complete this assessment, a member of their family may answer the questions on their behalf.

This will complete the patient's participation in the trial. With the participant's permission, the researchers at the recruiting hospital will contact the participant's family doctor (GP), Consultant and any other Health Care Professional involved in their care to let them know of the patient's participation in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with spontaneous, non-traumatic, supratentorial ICH with no underlying macrovascular or neoplastic cause admitted to a participating centre within 8 hours of symptom onset.
2. No concomitant health problems that, in the opinion of the principle Investigator (PI) or designee, would interfere with participation, administration of study drug or assessment of outcomes including safety.
3. Willing and able to give informed consent or consent available from a patient representative for trial inclusion including agreement in principle to receive study drug and undergo all study assessments.
4. Male or female aged 18 years or above.

Exclusion Criteria:

1. Severe ICH, unlikely to survive to 72 hours scan, in the opinion of the treating clinician. For example, a GCS score < 6 at time of consent);
2. Confirmed or suspected structural abnormality as cause of ICH (including tumour, vascular malformation).
3. Confirmed or suspected haemorrhagic transformation of an arterial or venous infarct.
4. Acute neurosurgery planned within 72 hours of admission.
5. Known active tuberculosis or active hepatitis.
6. Known active malignancy.
7. Neutropenia (absolute neutrophil count (ANC) <1.5 x10^9/L).
8. Abnormal renal function (creatinine clearance or estimated Glomerular Filtration Rate (eGFR) < 30 ml/minute) documented in the last 3 months prior to this ICH.
9. Live vaccinations within the last 10 days prior to this ICH.
10. Previous or concurrent treatment with IL-1Ra known at the time of trial entry or previous participation in this trial.
11. Previous or current treatment with etanercept or any other tumour necrosis factor alpha (TNFα) antagonist.
12. Known to have participated in a clinical trial of an investigational agent or device in the 30 days prior to symptom onset.
13. Known to have participated in a clinical trial of an investigational agent or device within 5 half-lives (of the previous agent or device) prior to symptom onset.
14. Known to be pregnant or breast-feeding or inability to reliably confirm that the patient is not pregnant.
15. Known diagnosis of Still's disease.
16. Clinically significant serious concurrent medical condition, premorbid illnesses, or concurrent serious infection, at the PI's (or designee's) discretion, which could affect the safety or tolerability of the intervention.
17. Known allergy to IL-1Ra or any of the excipients listed in the drug summary of product characteristics (SmPC).
18. Known allergy to other products that are produced by DNA technology using the micro-organism E. coli (e.g. E.coli derived protein).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Oedema extension distance (OED) | 72 hours (+/-12 hours) post symptoms onset
  Perihaematomal OED on CT scan at 72 hours (+/-12 hours), which equates to the average distance that oedema extends beyond the haematoma border.

SECONDARY OUTCOMES:
Early haematoma growth | between baseline and 72 hours post symptoms onset
  Early haematoma growth (defined as ≥33% or ≥6 ml increase in haematoma volume between baseline and 72 hours)
Early Neurological Decline (END) | between baseline and 72 hours post symptoms onset
  The average decrease of ≥2 in the Glasgow Coma Scale (GCS) score or an increase in the National Institutes of Health Stroke Scale (NIHSS) score ≥ 4, lasting longer than 8 h, requiring surgical intervention, or resulting in death.
Inflammatory markers | from day 0 (baseline) to day 4 post randomisation
  Area under the curve for inflammatory markers of C-reactive protein (CRP) versus Interleukin-6 (IL-6)
Quantitative blood-brain barrier permeability | day 2-4 post randomisation
  Measure of the blood-brain barrier permeability in the perihaematomal brain using a tracer kinetic model, which generates maps of the blood-brain transfer constant K^trans
modified Rankin Score (mRS) | 3 months post randomisation
  Measure of ordinal shift in degree of disability or dependence in daily activities
Stroke Impact Scale (SIS) | 3 months post randomisation
  stroke-specific quality of life measure
Fatigue severity score (FSS) | 3 months post randomisation
  Severity of fatigue and it's effect on the participant's activities and lifestyle
EQ-5D-5L | 3 months post randomisation
  health-related quality of life measure
Hospital Anxiety and Depression Scale (HADS) | 3 months post randomisation
  Measurement of mood

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Parry-Jones, PhD, MRCP, Principal Investigator — University of Manchester
Locations (1):
- Salford Royal NHS Foundation Trust, Manchester, North West, United Kingdom

REFERENCES:
- [Derived] Parry-Jones AR, Stocking K, MacLeod MJ, Clarke B, Werring DJ, Muir KW, Vail A. Phase II randomised, placebo-controlled, clinical trial of interleukin-1 receptor antagonist in intracerebral haemorrhage: BLOcking the Cytokine IL-1 in ICH (BLOC-ICH). Eur Stroke J. 2023 Sep;8(3):819-827. doi: 10.1177/23969873231185208. Epub 2023 Jul 15. PMID 37452707